CLINICAL TRIAL: NCT00592176
Title: The Effect of Bevacizumab (Avastin) on Pterygium
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F070323011
Record Dates: First submitted 2007-12-26; First posted 2008-01-11 (Estimated); Results first posted 2012-06-25 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2012-05

CONDITIONS: Pterygium
MeSH Terms: conditions — Pterygium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bevacizumab (Experimental): Bevacizumab injection: 0.1ml, 6 monthly doses plus baseline and 1 week post baseline
  Interventions: Drug: local injection of bevacizumab

INTERVENTIONS:
Drug: local injection of bevacizumab — Upon enrollment into the study: - initial injection of bevacizumab, a 1 week post-injection visit,and monthly visits thereafter for a total of 6 months. At the 1-month and 3-month visit post-injection visit, an additional bevacizumab injection will be offered if pterygium regression has not occurred. All injections of bevacizumab will consist of injecting 0.1mL of a 2.5mg/0.1mL concentration of bevacizumab into the head of the pterygium.

SUMMARY:
The purpose of this study is to determine whether local injection of bevacizumab might halt and or cause regression of pterygium growth. This may enable earlier treatment and prevention of pterygium growth into the patient's line of sight thereby limiting the need for surgery and improving quality of life for patients with pterygia.

ELIGIBILITY:
Inclusion Criteria:

* 19 years of age and older
* Diagnosis of pterygia
* healthy enough to make scheduled follow-up visits

Exclusion Criteria:

* Women of childbearing potential and males who plan to father a child during their participation in the study will be excluded from the study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2007-08; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tyler A Hall, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Callahan Eye Foundation Hospital, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab: The participants received an initial 0.5mL subconjunctival injection of bevacizumab(2.5mg/mL) beneath the pterygium at the limbus and again every month for a total of 3 injections.
Period: Overall Study
Arm/Group | Bevacizumab
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Bevacizumab
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: The Area the Pterygium Enlarged or Regressed as Measured From the Limbus Before and After Subconjunctival Bevacizumab Injection.
Description: Growth of the pterygium was defined as an increase in the area of the pterygium as measured from the limbus toward the visual axis. This would be a positive change value indicating progression
  Regression of the pterygium was defined as a decrease in the area of the pterygium length measured from the limbus toward the visual axis. This would be negative change value indicating regression.
Time Frame: Baseline and 3 months
Population: All subjects enrolled were analzyed.
Measure: Mean (Standard Deviation); unit: area in millimeters squared
Groups:
- Bevacizumab: Patients receiving bevacizumab treatment.
Arm/Group | Bevacizumab
Number analyzed (Participants) | 5
area in millimeters squared | 5.75 (2.91)
Statistical Analysis 1: Comparison: Bevacizumab; Test type: Superiority or Other; p = 0.83, t-test, 2 sided

2. Secondary Outcome: Number of Patients Having Surgical Removal of Pterygium.
Description: The number of patients having surgical removal of pterygium within 12 months.
Time Frame: 12 months
Population: All subjects enrolled were analzyed.
Measure: Number; unit: Participants
Arm/Group | Bevacizumab
Number analyzed (Participants) | 5
Participants | 0

ADVERSE EVENTS:
Arm/Group | Bevacizumab
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 4/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab (N=5)
Pulling at site of injection of avastin (Eye disorders) | 2 (2)
Subconjunctival hemorrhage at injection site (Eye disorders) | 1 (1)
Ocular Irritation (Eye disorders) | 1 (1) — Patient complained of irritation at site of injection which resolved.

LIMITATIONS AND CAVEATS:
Initially we aimed for 10 to 15 subjects but only enrolled 5 subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No